CLINICAL TRIAL: NCT01983475
Title: The Efficacy of Denosumab to Reduce Osteoporosis After Spinal Cord Injury
Brief Title: Denosumab Administration After Spinal Cord Injury
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: James J. Peters Veterans Affairs Medical Center (U.S. Federal Agency)
Collaborators: Kessler Institute for Rehabilitation (Industry)
Responsible Party: Principal Investigator, William A. Bauman, M.D., Director VA RR&D Center of Excellence for the Medical Consequences of SCI, James J. Peters Veterans Affairs Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 113536
Record Dates: First submitted 2013-11-06; First posted 2013-11-14 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Osteoporosis; Spinal Cord Injury
Keywords: Spinal Cord Injury; Denosumab; Osteoporosis; Dual Energy X-ray Absorptiometry
MeSH Terms: conditions — Osteoporosis; Spinal Cord Injuries | interventions — Denosumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): A group of participants will be randomized to the placebo group and will receive the identical volume of normal saline at parallel time points.
  Interventions: Drug: Placebo (identical Denosumab volume of normal saline)
- Denosumab (Experimental): A group of participants will be randomized to the experimental group and will have Denosumab (Prolia, 60 mg SC) administered at baseline, 6 and 12 months.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Denosumab — In clinical trials, denosumab (Amgen Inc., Thousand Oaks, CA), has been shown to be more potent in reducing osteoclastosis and function than bisphosphonates.39,40 The rate of bone loss in the lower extremity at sites of interest in patients with acute SCI has been reported to be several-fold greater than the rate of bone loss in postmenopausal women not prescribed antiresorptive medications, which is about 3-5% per year.11,50,51 The dose of denosumab chosen for our protocol in patients after acute SCI will be the same dose that has been shown to be efficacious to treat postmenopausal osteoporosis (60 mg SQ q 6 months).
  Other Names: Prolia
  Arms: Denosumab
Drug: Placebo (identical Denosumab volume of normal saline) — The placebo group will receive the identical volume of normal saline at parallel time points.
  Other Names: Unknown at this time
  Arms: Placebo

SUMMARY:
Sublesional bone loss after acute spinal cord injury (SCI) is sudden, progressive, and dramatic. After depletion of bone mass and the loss of architectural integrity, it may be difficult, if even possible, to restore skeletal mass and strength. Denosumab is a relative new, highly potent anti-resorptive agent that has proven efficacy in postmenopausal osteoporosis to improve bone mass and in solid tumor patients to prevent a skeletal-related event to a greater extent than that with bisphosphonate administration. In persons with complete motor lesions, bisphosphonates have not been effective at reducing bone loss at the knee, the site of greatest relevance because of its increased risk of fracture. Anti-RANKL therapy appears to be more potent than bisphosphonates in animal models of bone loss due to immobilization, suggesting that treatment with denosumab may prove to be an efficacious therapy for persons with acute SCI to preserve bone mass and strength.

DETAILED DESCRIPTION:
The primary objective of this study is to test the efficacy of a potent anti-resorptive agent, denosumab [receptor activator of nuclear factor-κB ligand (RANKL) antibody; Amgen Inc.] to preserve bone mass at the hip and knee and trabecular connectivity at the knee after acute SCI. Setting: patient enrollment, study drug administration and DXA scanning will be completed at the Kessler Institute for Rehabilitation (KIR) and pQCT measurements will be performed at Columbia University. A Randomized, double-blind, placebo-controlled parallel group trial.

Twenty-four subjects with acute, motor complete SCI (≤12 weeks) who have been admitted to the Kessler Institute for Rehabilitation (KIR) will be recruited for participation. The age of study participation will be males between the ages of 18 and 65 years old and females between the ages of 18 and 50 years old. Primary outcome measure will be BMD as measured by DXA and microarchitecture as measured by pQCT at the hip and knee.

ELIGIBILITY:
Inclusion Criteria:

1. Complete motor SCI [American Spinal Injury Association Impairment Scale (AIS) grade A and B];
2. Duration of injury <12 weeks; and
3. Males between the ages of 18 and 65 years old and females between the ages of 18 and 50 years old.

Exclusion Criteria:

1. Extensive life-threatening injuries in addition to SCI;
2. Acute fracture or extensive bone trauma;
3. History of prior bone disease (Paget's hyperparathyroidism, osteoporosis, etc.)
4. Post menopausal women;
5. Men with known hypogonadism prior to SCI;
6. Anabolic or Steroid hormonal therapy; within the past year and longer than six months;
7. Hyperthyroidism;
8. Cushing's disease or syndrome;
9. Severe underlying chronic disease;
10. Heterotopic ossification of the knee region (HO limited to the hip region only will not exclude subject participation);
11. History of chronic alcohol abuse;
12. Diagnosis of Hypocalcemia;
13. Pregnancy;
14. Existing dental condition/dental infection
15. Any patient taking a bisphosphonate for heterotopic ossification (HO);
16. Current diagnosis of cancer or history of cancer; and
17. Any patient receiving moderate or high dose corticosteroids (>40 mg/d prednisone or an equivalent dose of other corticosteroid) for longer than one week, not including drug administered in an attempt to preserve neurological function at the time of acute SCI.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-01; Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Bone mineral density (BMD) of the distal femur | Baseline, 1, 3, 6, 12, and 18 months after Denosumab administration
  Change in BMD at the distal femur will be obtained by dual energy X-ray absorptiometry (DXA) at baseline, 1, 3, 6, 12, and 18 months after Denosumab administration.

SECONDARY OUTCOMES:
Bone microarchitecture of the distal femur and proximal tibia. | Baseline, 12, and 18 months after Denosumab administration
  Change in microarchitecture at the distal femur and proximal tibia will be obtained by peripheral quantitative computerized tomography (pQCT) at baseline, 12, and 18 months after Denosumab administration.

CONTACTS AND LOCATIONS:
Overall Officials: William A Bauman, M.D., Principal Investigator — James J. Peters VA Medical Center; Steven C Kirshblum, M.D., Principal Investigator — Kessler Institute for Rehabilitation
Locations (2):
- United States (2):
  - Kessler Institute for Rehabilitation, West Orange, New Jersey
  - James J. Peters VA Medical Center, The Bronx, New York

REFERENCES:
- [Background] Reid IR, Miller PD, Brown JP, Kendler DL, Fahrleitner-Pammer A, Valter I, Maasalu K, Bolognese MA, Woodson G, Bone H, Ding B, Wagman RB, San Martin J, Ominsky MS, Dempster DW; Denosumab Phase 3 Bone Histology Study Group. Effects of denosumab on bone histomorphometry: the FREEDOM and STAND studies. J Bone Miner Res. 2010 Oct;25(10):2256-65. doi: 10.1002/jbmr.149. PMID 20533525
- [Background] Kendler DL, Roux C, Benhamou CL, Brown JP, Lillestol M, Siddhanti S, Man HS, San Martin J, Bone HG. Effects of denosumab on bone mineral density and bone turnover in postmenopausal women transitioning from alendronate therapy. J Bone Miner Res. 2010 Jan;25(1):72-81. doi: 10.1359/jbmr.090716. PMID 19594293
- See also: Spinal Cord Damage Research Center — http://www.scirc.org/